CLINICAL TRIAL: NCT06473857
Title: Design, Implementation and Evaluation of an Intervention Within an Online Community Game for the Development of Mental Health Literacy in Adolescents and Young Adults
Brief Title: Design, Implementation and Evaluation of an Intervention Within Video Game for Mental Health Literacy in Adolescents and Young Adults
Acronym: SCOTT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A21024HS; CNAM_SCOTT_CIC1426_alberti (Other: CNAM)
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Literacy
Keywords: mental health; literacy; adolescent and young adults; video games
MeSH Terms: conditions — Psychological Well-Being; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health Literacy intervention (Experimental): Mental health literacy interventions delivered online for adolescents and young adults on, 3 modalities : webconferences, build battle, serious games
  Interventions: Behavioral: Mental health literacy intervention
- Other topic intervention - not related to mental health (Other): Other topics online interventions for adolescents and young adults, 3 modalities : webconferences, build battle, serious games
  Interventions: Behavioral: Non mental health intervention

INTERVENTIONS:
Behavioral: Mental health literacy intervention — Online interventions for adolescents and young adults on mental health literacy, 3 modalities : webconferences, build battle, serious games
  Arms: Mental Health Literacy intervention
Behavioral: Non mental health intervention — Online interventions for adolescents and young adults on other topics, 3 modalities : webconferences, build battle, serious games
  Arms: Other topic intervention - not related to mental health

SUMMARY:
Context Adolescence and early adulthood are crucial periods for the development and maintenance of habits, behaviors and beliefs favorable to health and mental well-being. These can have significant lifelong health consequences and social costs. In this age group, the Internet and smartphones are predominant. Based on these two observations, the project proposes to use the Internet, and more specifically, an online game, as a vector for public health intervention. Health literacy is recognized as a key determinant of health. It refers to the motivation and skills of individuals to access, understand, evaluate and use information to make decisions about their health. Improving the level of literacy is a major public health challenge if the population is to be in a position to take better charge of its health, particularly its mental health.

Objective To evaluate the effect of a public health intervention on the development of mental health literacy in adolescents and young adults (15-25 years) delivered within an existing online community game.

Research hypothesis Developing and delivering a (multicomponent) public health intervention in an original setting, such as the game Minecraft, to a community of adolescents and young adults will improve their mental health literacy and thus enhance the primary, secondary and tertiary prevention of mental health disorders.

Methods The project's overall methodology is based on a multidisciplinary approach. A pilot phase has already enabled us to develop the theoretical framework and constituent elements of an intervention, as well as its acceptability and feasibility.

Intervention We will conduct a pragmatic cohort multiple randomised controlled trial over 24 months. The chosen methodology will enable us to implement an intervention with different components.

The intervention will involve: collective challenges of various kinds (component A) and exchanges with influencers of different profiles (component B). The control group will be offered access to conventional sources of health information and ""placebos"" of the components described above. The theme is mental health literacy, and the intervention delivered will equip the players (capacity-building, recognizing ill-being, warning signs, resources, etc.) to ultimately enable them to react better (empowerment) and thus promote young people's mental health.

Evaluation The evaluation will follow the Medical Research Council's recommendations for the evaluation of complex interventions. It will consist of a process evaluation and an evaluation of effectiveness, all of which will be based on the use of mixed methods (observations of players receiving the intervention, analysis of chat exchanges made by players during the intervention, evaluation questionnaires and a standardized grid for collecting process indicators). The primary endpoint for the effect analysis is the mental health literacy score (global score) measured by the MHLq including four dimensions: (1) knowledge of mental health problems; (2) mistaken beliefs/stereotypes; (3) help-seeking and first-aid skills; and (4) self-help strategies.

Perspectives The results of this research project will make it possible to 1) develop new relevant interventions on various health topics, using the results obtained for the different interventions carried out within Minecraft 2) Contribute to the evidence base on the effectiveness of Internet-based interventions.

DETAILED DESCRIPTION:
Context Adolescence and early adulthood are crucial periods for the development and maintenance of habits, behaviors and beliefs favorable to health and mental well-being. These can have significant lifelong health consequences and social costs. In this age group, the Internet and smartphones are predominant. Based on these two observations, the project proposes to use the Internet, and more specifically, an online game, as a vector for public health intervention. Health literacy is recognized as a key determinant of health. It refers to the motivation and skills of individuals to access, understand, evaluate and use information to make decisions about their health. Improving the level of literacy is a major public health challenge if the population is to be in a position to take better charge of its health, particularly its mental health.

Objective To evaluate the effect of a public health intervention on the development of mental health literacy in adolescents and young adults (15-25 years) delivered within an existing online community game.

Research hypothesis Developing and delivering a (multicomponent) public health intervention in an original setting, such as the game Minecraft, to a community of adolescents and young adults will improve their mental health literacy and thus enhance the primary, secondary and tertiary prevention of mental health disorders.

Methods The project's overall methodology is based on a multidisciplinary approach. A pilot phase has already enabled us to develop the theoretical framework and constituent elements of an intervention, as well as its acceptability and feasibility.

Intervention We will conduct a pragmatic cohort multiple randomised controlled trial over 24 months. The chosen methodology will enable us to implement an intervention with different components.

The intervention will involve: collective challenges of various kinds (component A) and exchanges with influencers of different profiles (component B). The control group will be offered access to conventional sources of health information and ""placebos"" of the components described above. The theme is mental health literacy, and the intervention delivered will equip the players (capacity-building, recognizing ill-being, warning signs, resources, etc.) to ultimately enable them to react better (empowerment) and thus promote young people's mental health.

Evaluation The evaluation will follow the Medical Research Council's recommendations for the evaluation of complex interventions. It will consist of a process evaluation and an evaluation of effectiveness, all of which will be based on the use of mixed methods (observations of players receiving the intervention, analysis of chat exchanges made by players during the intervention, evaluation questionnaires and a standardized grid for collecting process indicators). The primary endpoint for the effect analysis is the mental health literacy score (global score) measured by the MHLq including four dimensions: (1) knowledge of mental health problems; (2) mistaken beliefs/stereotypes; (3) help-seeking and first-aid skills; and (4) self-help strategies.

Perspectives The results of this research project will make it possible to 1) develop new relevant interventions on various health topics, using the results obtained for the different interventions carried out within Minecraft 2) Contribute to the evidence base on the effectiveness of Internet-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* French speaking Minecraft players (15 to 25 years old)

Exclusion Criteria:

-

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
MHLq : the mental health literacy questionnaire for young adults | 2 months
  Measure of the variation in the mental health literacy questionnaire score among young adults before and 2 months after an online intervention on mental health literacy

CONTACTS AND LOCATIONS:
Overall Officials: Enora LE ROUX, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Robert Debré, Paris, France